CLINICAL TRIAL: NCT06770348
Title: Exploring the Origin of Consciousness Through Disorders of Consciousness: a PET Study"
Brief Title: Investigating the Localization of Consciousness Through Patients with Disorders of Consciousness: Anterior Vs. Posterior Cortex Debate
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Anqi Wang, Principal Investigator, Hangzhou Normal University
Other Study IDs: 20230630
Record Dates: First submitted 2024-12-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Disorders of Consciousness
Keywords: disorders of consciousness; MCS; PET; UWS
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- UWS (Unresponsive Wakefulness Syndrome): presence of basic arousal, localization to sound, auditory startle responses, visual startle responses, flexion withdrawal, abnormal posturing, vocalization/oromotor responses, and/or reflexive oromotor movements.
- MCS (Minimally Conscious State): based on the following criteria: stable responses to commands, the ability to repeat commands, object recognition, understandable speech, incomplete communication, object localization, visual tracking, visual object localization, voluntary motor responses, manipulation of objects, and/or localization of noxious stimuli.
- HC (Healthy control): people with full consciousness

SUMMARY:
Patients enrolled in the study underwent five assessments using the CRS-R(Coma Recovery Scale-Revised) within 10 days, along with an 18F-FDG-PET scan.

DETAILED DESCRIPTION:
Patients enrolled in the study underwent five assessments using the CRS-R (Coma Recovery Scale-Revised) within 10 days, along with an 18F-FDG-PET (18F-fluorodeoxyglucose-positron emission tomography) scan. The CRS-R evaluations were conducted by professionally trained and highly experienced personnel. During the CRS-R assessments, patients' behavioral responses were recorded in the domains of visual, auditory, motor, oromotor/verbal, communication, and arousal. Based on the optimal CRS-R results obtained within the 10-day period, patients were categorized into MCS (Minimally consciousness state, criteria: consistent command-following, reproducible responses to commands, object recognition, intelligible verbalization, partially accurate communication, object localization, visual pursuit and visual object localization, spontaneous motor responses, object manipulation, and/or localization to noxious stimulation) or UWS (Unresponsive wakefulness syndrome, criteria: preserved wakefulness accompanied by behavioral responses such as localization to sound, auditory startle, visual startle, withdrawal/flexion movements, abnormal posturing, vocalizations/oromotor movements, and reflexive oromotor responses). All patients exhibited stable vital signs. For data analysis, a healthy control group from Belgium was included to compare brain metabolism between patients with disorders of consciousness and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of disorders of consciousness after 5 CRS-R assessments;
* Age >18 years;
* Stable vital signs;
* No use of sedatives or neuromuscular blockers within 24 hours prior to enrollment.

Exclusion Criteria:

* Acute-phase patients (injury duration <28 days);
* Fewer than 5 CRS-R assessments completed within 10 days;
* Patients diagnosed with EMCS (Emerging Minimally Conscious State);
* Patients with unclear diagnoses (cases where experienced evaluators could not reach a consensus diagnosis);
* Patients with persistent seizures.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The enrolled patients were from Shanghai Yongci Rehabilitation Hospital, The Second People's Hospital of Hefei , and the First Affiliated Hospital, Zhejiang University school of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Brain metabolism in patients with disorders of consciousness was measured by 18F-FDG-PET | From enrollment to the end of CRS-R assessment in 10 days
  Patients were assessed using the CRS-R (Coma Recovery Scale-Revised) five times within 10 days, and an 18F-FDG-PET scan was performed. The assessors for the CRS-R evaluations were professionally trained and highly experienced. During the CRS-R assessment, the patients' behavioral performance in the areas of visual, auditory, motor, oromotor/speech, communication, and arousal were recorded. The patient's best CRS-R assessment score within the 10-day period was used to classify them into MCS (Minimally Conscious State) and UWS (Unresponsive Wakefulness Syndrome).

CONTACTS AND LOCATIONS:
Locations (1):
- The enrolled patients were from Shanghai Yongci Rehabilitation Hospital, The Second People's Hospital of Hefei , and the First Affiliated Hospital, Zhejiang University school of Medicine., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided